CLINICAL TRIAL: NCT07334457
Title: Study of Platelet Population Changes Under Circulatory Support With ECMO
Acronym: ECMO-POP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9614
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Failure; Respiratory Failure
Keywords: Cardiac Failure; Respiratory Failure
MeSH Terms: conditions — Heart Failure; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Advances in flow cytometry techniques have led to a better understanding of platelet phenotypes and have revealed the existence of four major platelet populations with distinct functional properties (native, proaggregating, procoagulating, or apoptotic). These phenotypes have a significant impact on the hemostatic capacity of blood platelets, and a proportional change in these populations during ECMO treatment could, at least in part, contribute to the observed complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years) treated in one of the intensive care units of the Anesthesia and Intensive Care Department at Strasbourg University Hospital.
* Implanted with veno-arterial or veno-venous ECMO within the previous 24 hours.

Exclusion Criteria:

* Subject who has expressed their opposition to participating in the study.
* Subject under legal protection.
* Subject under guardianship or curatorship.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - Adult patient (≥18 years) treated in one of the intensive care units of the Anesthesia and Intensive Care Department at Strasbourg University Hospital and implanted with veno-arterial or veno-venous ECMO within the previous 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03-11 (Estimated)

PRIMARY OUTCOMES:
Proportional Changes in the Different Platelet Populations (native, proaggregating, procoagulant, or apoptotic) | Days 1, 3, and 7 after the initiation of ECMO treatment.
  Proportional Changes in the Different Platelet Populations (native, proaggregating, procoagulant, or apoptotic) on Days 1, 3, and 7 after the initiation of ECMO treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'anesthésie-réanimation - CHU de Strasbourg - France, Strasbourg, France